CLINICAL TRIAL: NCT05462639
Title: ELRANATAMAB (PF-06863135) MONOTHERAPY EXPANDED ACCESS PROTOCOL FOR TREATMENT OF PATIENTS WITH RELAPSED/REFRACTORY MULTIPLE MYELOMA WHO ARE REFRACTORY TO AT LEAST ONE PROTEASOME INHIBITOR, ONE IMMUNOMODULATORY DRUG AND ONE ANTI-CD38 ANTIBODY AND HAVE NO ACCESS TO OTHER COMPARABLE/ALTERNATIVE THERAPY
Brief Title: Elranatamab Expanded Access Protocol in Adults With Relapsed/Refractory Multiple Myeloma
Acronym: MAGNETISMM17
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071017
Record Dates: First submitted 2022-06-20; First posted 2022-07-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Erlanatamab; Expanded Access; MM17; MagnetisMM-17; BCMA; BCMA antibody; Advanced multiple myeloma; Relapse/Refractory; RRMM; MagnetisMM; MagnetisMM US; Bispecific Antibody
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Elranatamab (PF-06863135) — BCMA-CD3 bispecific antibody

SUMMARY:
Elranatamab is a bispecific antibody: binding of elranatamab to CD3- expressing T-cell and BCMA- expressing multiple myeloma cells causes targeted T-cell mediated cytotoxicity.

This expanded access protocol will provide access to elranatamab until it becomes commercially accessible to patients who are refractory to at least one proteasome inhibitor, one immunomodulatory drug and one anti-CD38 antibody and have no access to other comparable/alternative therapy and for whom elranatamab could be a possible treatment option.

DETAILED DESCRIPTION:
Study C1071017 is a single-arm, open-label study in patient with relapsed /refractory multiple myeloma.

Each patient will receive study intervention until disease progression, unacceptable toxicity, withdrawal of consent, study termination or until elranatamab becomes commercially accessible.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of MM as defined according to IMWG criteria .
* Patients who are ineligible for participation in any ongoing clinical trial of elranatamab, including lack of access due to geographical limitations, and who have exhausted all other treatment options or experience lack of access to commercially available therapies due to geographical, financial or socioeconomic limitations.
* Measurable disease at screening based on IMWG criteria as defined by at least 1 of the following:
* Serum M-protein ≥0.5 g/dL (≥5 g/L)
* Urinary M-protein excretion ≥200 mg/24 hours
* Involved FLC ≥10 mg/dL (≥100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FLC ratio (<0.26 or >1.65).
* Refractory to at least one IMiD, one PI, and one anti-CD38 antibody.
* Relapsed/refractory to last anti-MM regimen.
* ECOG performance status 0-1.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1.
* Not pregnant, willing to use contraception

Exclusion Criteria:

* Smoldering MM; plasma cell leukemia; POEMS syndrome; Waldenström's macroglobulinemia; amyloidosis; stem cell transplant within 12 weeks prior to enrollment or active GVHD
* Previous treatment with BCMA directed therapy;
* Active HBV, HCV, SARS- CoV-2, HIV or any active, uncontrolled bacterial, fungal, or viral infection.

Active infections must be resolved at least 14 days prior to enrollment.

* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ or Stage 0/1 with minimal risk of recurrence per treating physician.
* Previous administration with an investigational drug or vaccine within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (30):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 120), Los Angeles, California
  - UC Irvine Health, Orange, California
  - UC Irvine Medical Center, Orange, California
  - Baptist Hospital of Miami, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Hospital West Laboratory Services, Pembroke Pines, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Franciscan Health, Indianapolis, Indiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - MSK Nassau, Uniondale, New York
  - OhioHealth Arthur G.H. Bing, MD Cancer Center, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Baylor Scott & White Charles A. Sammons Cancer Center, Dallas, Texas
  - Baylor University Medical Center, Investigational Drug Services, Department of Pharmacy, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Texas Oncology, Dallas, Texas
- Canada (3):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071017